CLINICAL TRIAL: NCT06633107
Title: The Impact of Cardiac Rehabilitation Exercise Therapy on the Quality of Life of Patients With Chronic Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AMCIIT240908; B202437 (Other Grant/Funding Number: Chongqing Administration of Sport)
Record Dates: First submitted 2024-09-26; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Medically relevant pharmacotherapy combined with rehabilitation exercise therapy. Continued rehabilitation exercise therapy intervention 3 months after discharge.
  Interventions: Behavioral: Cardiac、rehabilitation、exercise
- control group (No Intervention): Only medically relevant medications are given during hospitalization. No rehabilitation exercise therapy intervention for 3 months after discharge.

INTERVENTIONS:
Behavioral: Cardiac、rehabilitation、exercise — Routine cardiac rehabilitation treatment + corresponding rehabilitation exercise therapy prescription according to the condition: (1) slow walking + stairs climbing + standing aerobic exercise for patients with cardiac function level I; Grade II patients should take slow walking + standing aerobics; Grade III patients undergo bedside chair aerobics; Class IV aerobic exercises on bed.
  After discharge aerobic exercise with the help of community exercise equipment. The duration is gradually increased from 10-20min to 30-40min each time; Gradually increase the intensity from 55% to 60% of the maximum heart rate and not exceed 85% (maximum heart rate (times / min) = 220 - age (years)); The frequency gradually increased from 3 days/week to 5 days/week
  Arms: experimental group

SUMMARY:
This study aims to explore the effectiveness of cardiac rehabilitation exercise therapy in improving the quality of life of patients with chronic heart failure during hospitalization and after discharge. The specific research content includes screening patients who meet the diagnosis of "chronic heart failure" among cardiovascular inpatients from October 2024 to October 2025. Among these patients, those who meet the inclusion criteria and can participate in the study for more than three months are selected. After a detailed explanation, they sign an informed consent form. Finally, eligible patients are included in the study and divided into a control group and an observation group using a random number table method. Various indicators of the enrolled patients are monitored and recorded, including: general information (gender, age, height, weight, BMI, etc.) Educational background, medical history, medication history, laboratory test results, 6-minute walk test results, New York Heart Association (NYHA) cardiac function grading, ultrasound examination results, Minnesota Heart Failure Quality of Life Scale, 1-year mortality assessment for heart failure patients, and prognosis evaluation for chronic heart failure patients. Patients in the control group received routine cardiac rehabilitation guidance; Patients in the observation group receive routine cardiac rehabilitation guidance and develop corresponding rehabilitation exercise therapy prescriptions based on their condition: ① Patients with heart function level I perform slow walking, climbing stairs, and standing aerobic exercises; Grade II patients undergo slow walking and standing aerobic exercises; Grade III patients perform aerobic exercises on bedside seats; Grade IV aerobic exercise on the bed. Guide and supervise two groups of patients to engage in rehabilitation exercises during hospitalization, and record the required indicators during exercise. After discharge, the patient will be followed up for a period of three months. The rehabilitation exercise data will be accurately and completely recorded in the form of a diary by the patient and/or family members, and feedback will be provided weekly, including time, location, exercise time, exercise method, heart rate, and other data. Guidance on home rehabilitation exercise therapy for the observation group: ① Warm up exercise for 5-10 minutes (to awaken the body through warm-up exercise and reduce strains during exercise). Choose the warm-up exercise method according to your own situation, including "chest expansion exercise, dynamic back extension, standing shoulder activation, foot wrap around the" 8 "shape, knee joint warm-up, standing lateral flexion, full body stretching, relaxation jumping, slow jogging in place, and continuous knee strikes" Aerobic exercise with the help of community sports equipment. The duration gradually increased from 10-20 minutes each time to 30-40 minutes; The intensity gradually increases from 55% maximum heart rate to 60%, not exceeding 85% (maximum heart rate (beats/minute)=220- age (years)); The frequency gradually increased from 3 days/week to 5 days/week; Sports equipment can be selected based on community equipment, such as elliptical machines, Tai Chi massagers, cycling machines, spacewalkers, treadmills, etc Rest (if discomfort occurs during exercise, immediately stop exercising and rest in place). This study used experimental and observational methods to analyze and evaluate various indicator data at admission, discharge, and 3 months of home rehabilitation. Ultimately, it was concluded that cardiac rehabilitation exercise therapy is effective and worthy of promotion in improving the quality of life of patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic heart failure
* NYHA classification of cardiac function of class I. II. III.IV.
* Must be able to complete the training

Exclusion Criteria:

* Cognitive impairment
* Impairment of physical mobility

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
New York Heart Association (NYHA) Classification of Cardiac Function | The first day of hospitalized;The last day of hospitalized;Through study completion, an average of 3 months
  Class I.II. III. IV.

SECONDARY OUTCOMES:
NT-proBNP | The first day of hospitalized;The last day of hospitalized;Through study completion, an average of 3 months
  Overall standard: The normal value is less than 300 ng / L. Age stratification: < 50 years: NT-probnp levels greater than 450 ng / L may indicate acute heart failure. 50-75 years: NT-probnp levels greater than 900 ng / L may indicate acute heart failure. Age 75 and older: NT-probnp levels greater than 1800 ng/ L may indicate acute heart failure. NT-probnp > 1200 ng / L may indicate acute heart failure if the patient has renal insufficiency (eg, GFR < 60 ml/ min).
6-minute walking experiment（6MWT） | The first day of hospitalized;The last day of hospitalized;Through study completion, an average of 3 months
  Severe heart failure：6MWD is less than 150meters Moderate heart failure：6MWD is 150 to 450meters Mild heart failure：6MWD is more than 450meters
Minnesota Heart Failure Quality of Life Scale,MLHFQ | The first day of hospitalized;The last day of hospitalized;Through study completion, an average of 3 months
  The MLHFQ has 21 entries measuring the quality of life from three domains: the physical domain (entries 2, 3, 4, 5, 6, 7, 12, 13), the emotional domain (entries 17, 18, 19, 20, 21) and the other domains (entries 1, 8, 9, 10, 11, 14, 15, 16). Each MLHFQ entry is a 6-paragraph scoring method with 0-5 points. The original minimum score for each entry is 0 (best), the highest score is 5 (worst), and the total score for each entry is added up. As a result, the original combined score of 21 entries was 0 (best) to 105 (worst); The physical area scores are 0 (best) to 40 (worst), the emotional area scores is 0 (best), 25 (worst) and the other areas scores are zero (best) and 40 (worse). Higher scores indicate poorer quality of life, and lower scores mean better quality of life.
Ejection fraction | The first day of hospitalized;The last day of hospitalized;Through study completion, an average of 3 months
  Ejection fraction (EF) is the percentage of stroke output as a percentage of the ventricular end-diastolic volume. The normal value is 50-70%. Left ventricle ejection fraction (LVEF): Normal range: 55% -65%. Right ventricle ejection fraction: normal range: ≥ 40%.